CLINICAL TRIAL: NCT01471158
Title: Patient Preference Comparison of AZARGA Versus COSOPT After Single Doses in Patients With Open-Angled Glaucoma or Ocular Hypertension
Brief Title: Patient Preference Comparison of AZARGA Versus COSOPT in Patients With Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-09-18
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Glaucoma
Keywords: Primary open-angle glaucoma; ocular hypertension; pigment dispersion glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Azarga; dorzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azarga/Cosopt (Active Comparator): Following administration of the baseline dose (each intervention instilled in one eye in a contralateral fashion to establish baseline ocular comfort for each medication), Azarga will be instilled one drop in each eye on Day One, after which Cosopt will be administered one drop in each eye on Day Two.
  Interventions: Drug: Brinzolamide/Timolol Maleate Fixed Combination (AZARGA); Drug: Dorzolamide/timolol Maleate Fixed Combination (COSOPT)
- Cosopt/Azarga (Active Comparator): Following administration of the baseline dose (each intervention instilled in one eye in a contralateral fashion to establish baseline ocular comfort for each medication), Cosopt will be administered one drop in each eye on Day One, after which Azarga will be administered one drop in each eye on Day Two.
  Interventions: Drug: Brinzolamide/Timolol Maleate Fixed Combination (AZARGA); Drug: Dorzolamide/timolol Maleate Fixed Combination (COSOPT)

INTERVENTIONS:
Drug: Brinzolamide/Timolol Maleate Fixed Combination (AZARGA) — Brinzolamide/timolol maleate fixed combination, one drop instilled in one eye at baseline, followed by one drop instilled in each eye once in either first intervention period or second intervention period.
  Other Names: AZARGA®
Drug: Dorzolamide/timolol Maleate Fixed Combination (COSOPT) — Dorzolamide/timolol maleate fixed combination, one drop instilled in one eye at baseline, followed by one drop instilled in each eye once in either first intervention period or second intervention period.
  Other Names: COSOPT®

SUMMARY:
The purpose of this study is to assess patient preference of AZARGA® compared to COSOPT® after a single drop of each medication is administered to both eyes, in patients with open-angled glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, primary open-angle or pigment dispersion glaucoma in both eyes.
* On a stable regimen intraocular pressure (IOP) lowering medication within 30 days of screening visit.
* IOP considered to be safe (in the opinion of the investigator) in both eyes in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
* Willing to discontinue use of all other ocular drugs (prescribed and over-the-counter) prior to receiving the screening dose during Screening Visit and for the course of the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity, or poor tolerance to any component of the preparations to be used in this study that is deemed clinical significant in the opinion of the Principal Investigator.
* Corneal dystrophies in either eye.
* Risk of visual field or visual acuity worsening as a consequence of participating in this study, in the investigator's best judgment.
* Bronchial asthma or a history of bronchial asthma, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* History of severe allergic rhinitis.
* Participation in any other investigational study within 30 days prior to the Screening/Baseline Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Discomfort | One minute after instillation
  One drop of medication will be instilled in each eye. At one minute after instillation, subject will be given an Ocular Discomfort Scale and will record ocular discomfort on a questionnaire using a 10-point scale, with 0 being no discomfort and 09 being substantial discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Abayomi Ogundele, PharmD, Study Director — Alcon Research
Locations (1):
- Centro Oftalmológico, Buenos Aires, Argentina

REFERENCES:
- [Result] https://www.dovepress.com/preference-for-a-fixed-combination-of-brinzolamidetimolol-versus-dorzo-peer-reviewed-article-OPTH